CLINICAL TRIAL: NCT04888676
Title: Clinical Evaluation of Self- Adhesive Bulk-fill Resin Composite Versus Conventionally Bonded Bulk-fill Resin Composite in Restoration of Proximal Lesions Over a Period of 18 Months Follow-up: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Self- Adhesive Bulk-fill Resin Composite Versus Conventionally Bonded Bulk-fill Resin Composite in Restoration of Proximal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed mohamed sabry mohamed, Principal Investigator, Assistant lecturer at Conservative department., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: cons21
Record Dates: First submitted 2021-05-06; First posted 2021-05-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Dental Caries Class II

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Controlled Trial. Trial type: Two, Parallel arm design. Trial framework: Equivalence frame Allocation ratio: 1:1.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants Participants will be blinded to the technique used, since the patient will attend the same number of visits and he can not differentiate between different restorative materials.
  Blinding of the operator The operator cannot be blinded because of the use of different restorative materials applied in each group.
  The outcome assessor The outcome assessor will be blinded to the material used. This will be performed by M.A. and Y.H. Therefore it is necessary that the assessors won't be included in the preclinical assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self- Adhesive Bulk fill Resin Composite ( Surefil one™ ,Dentsupply Sirona) (Experimental): New Surefil one™ restorative Self-adhesive: no etching, bonding or cavity conditioning inserted in increments of up to 4 mm in thickness.
  Interventions: Procedure: Class II Restoration
- Bulkfill Resin Composite. (Tetric N-Ceram Bulk Fill ) (Active Comparator): after selective etching of enamel and bonding, the bulk-fill composite resins are inserted in increments of up to 4 mm in thickness.
  Interventions: Procedure: Class II Restoration

INTERVENTIONS:
Procedure: Class II Restoration — A Class II cavity will be prepared after local anesthesia has been given as required.Rubber dam isolation will be done.Sectional matricing and wedging will be done. Followed by, placement of restorative material according to the randomization sequence.followed by filling of cavity in increments of 3-4mm

SUMMARY:
This study will be conducted to evaluate and compare the clinical performance of Self- Adhesive Bulk fill Resin Composite Versus Conventionally Bonded Bulk fill resin composite in Restoration of Proximal Lesions Over a Period of 18 months Follow-up

Examination and selection of all patients will be done according to inclusion and exclusion criteria.A Class II cavity will be prepared after local anesthesia has been given as required. Sectional matricing and wedging will be done. Followed by, placement of restorative material according to the randomization sequence,. For the intervention: The sectional matrix will be applied first , followed by filling of cavity with Advanced Self- Adhesive bulk-fill Resin Composite. (Surefil one™ ,Dentsupply Sirona) in increments of 3-4mm,For the control group:

The sectional matrix will be applied first , followed by filling of cavity with bulk-fill resin composite material (GrandioSO x-tra® bulk) in increments of 3-4mm,Clinical evaluation will be done using using USPHS criteria at 6,12 and 18 months follow up.

DETAILED DESCRIPTION:
A) Participants, interventions & outcomes 9. Study setting Study will be conducted in the Conservative Dentistry Department, Faculty of Dentistry - Cairo University.

10. Eligibility criteria 10.a.1 Inclusion criteria:

Patient-related criteria:

* Patients consulting in one of the outpatient clinics listed above.
* Able to tolerate necessary restorative procedures.
* Provide informed consent.
* Accepts the 18 months follow-up period.

Tooth related criteria:

• Teeth with primary proximal carious lesions .

* Teeth are vital according to pulp-sensitivity tests. 10.a.2 Exclusion criteria

Patient-related criteria:

* Medically compromised patients, as they will not be able to attend multiple appointments or may require special management.
* Pregnant women; as radiographs cannot be taken for them.
* Allergy to any of the restorative materials, including anesthetics.
* Uncooperative patients, will not abide by the instructions or attend the appointments.

Tooth related criteria:

• Deciduous teeth; as the study is targeting only permanent teeth.

* Teeth with previous restorations, which may add another variable to the study (type of old restorative material, extent of recurrent caries).
* Spontaneous pain or prolonged pain after sensitivity tests (cold and electrical tests), which would indicate irreversible pulpal damage.
* Negative sensitivity tests, periapical radiolucencies and sensitivity to axial or lateral percussion, which would indicate pulp necrosis.
* Teeth presenting external or internal resorption, with adverse pulpal reactions which may affect the outcome of the study.
* Teeth with cervical caries; which can't be evaluated on periapical radiographs. 11. Interventions 11.a. Examination and diagnosis: Examination and selection of all patients will be done according to inclusion and exclusion criteria. Diagnosis of patients' chief complaint and teeth that will be involved in this study will be done. Teeth are to be chosen according to standardized radiographic examination. Teeth should have proximal, primary carious lesions .

  11.b. Cavity preparation procedure: A Class II cavity will be prepared after local anesthesia has been given as required. The cavity will be prepared using a high-speed hand-piece with air and water coolant and diamond burs of different sizes. Sharp excavators will allow accessible removal of soft carious lesions will be used. Any tooth that will suffer from pulpal exposure will be excluded from the study. Finishing of the cavity walls will be done using a fine-grit, yellow coded, diamond bur.

  11.c. Isolation: Rubber dam isolation will be done. 11.d. Matricing and wedging: Sectional matricing and wedging will be done. Followed by, placement of restorative material according to the randomization sequence.

  11.e. For the intervention: The sectional matrix will be applied first , followed by filling of cavity with Advanced Self- Adhesive bulk-fill Resin Composite. (Surefil one™ ,Dentsupply Sirona) in increments of 3-4mm, as required to end up with leaving an occlusal space on top of at least 2mm. Finally finishing and occlusal adjustment will be done under water spray by using superfine diamond burs. Polishing will be done using pre-impregnated rubber cups. Materials will be manipulated according to manufacturer instructions.

  11.f. For the control group: The sectional matrix will be applied first , followed by filling of cavity with bulk-fill resin composite material (GrandioSO x-tra® bulk) in increments of 3-4mm, as required to end up with leaving an occlusal space on top of at least 2mm. Finally finishing and occlusal adjustment will be done under water spray by using superfine diamond burs. Polishing will be done using pre-impregnated rubber cups. Materials will be manipulated according to manufacturer instructions.

  11.g. Intervention modification: Restoration will be removed when there are any signs of leakage, fracture or severe post-operative pain due to pulpal response.

  11.h. Intervention adherence: The patients' understanding of their conditions and treatments, and the amount of information given to the patient is positively related to adherence to the study and instructions given. Thus, the operator (M.S.) will inform the participants about all steps from the beginning to the end and explain the importance of restoring their teeth with such esthetic restorative materials, following instructions, attending follow up visits and how to maintain good oral hygiene. This will be done using simple oral conversation, emphasized by written and illustrated material whenever possible. Oral hygiene of the participants will be enhanced before intervention and any other chief and subsidiary complaint will be managed in order to modify their behavior.

  12. Outcomes: Clinical evaluation using USPHS criteria. 14. Sample Size : We are planning a study of independent cases and controls. Sample size was calculated based on the previous study by Guney et al in 2020. Prior data indicated that the probability of score A for marginal adaptation for bulk fill composite was 0.861 and score B was 0.139 with effect size w 0.722 (n=16). If the estimated probability of score A for marginal adaptation for self adhesive restorative material is 0.85 and score B is 0.15 with effect size w 0.7 (n=17), we will need to study a total of 33 restorations to be able to reject the null hypothesis that the success rates for case and controls are equal with probability (power) 0.8. This was increased to 40 subjects, 20 in each group to compensate for losses during follow up. The type I error probability associated with this test of this null hypothesis is 0.05. Sample size was calculated using G*Power version 3.1.9.2 for windows using chi-square test 15. Recruitment: Patients will be recruited by the principle investigator (M.S.) from outpatient clinic of conservative dentistry department in Faculty of Dentistry, Cairo University; from which eligible patients will be recruited to fulfill the eligibility criteria according to participant timeline.

B) Assignment of interventions 16. Allocation - sequence generation 16.a. Random sequence generation (Randomization): Simple randomization will be assigned for participants by generating numbers from 1:48 using Random Sequence Generator, Randomness and Integrity Services Ltd (https://www.random.org/) by D.K. . Each generated random number will represent assigning both intervention and comparator to each patient in a random manner.

16.b. Allocation concealment mechanism: The restorative technique will be selected according to randomized numbers in a sealed envelope.

16.c. Implementation: Randomization will be performed by D.K. 17. Blinding Double Blinded; The participants Participants will be blinded to the technique used, since the patient will attend the same number of visits and he can not differentiate between different restorative materials.

Blinding of the operator The operator cannot be blinded because of the use of different restorative materials applied in each group.

The outcome assessor The outcome assessor will be blinded to the material used. This will be performed by M.A. and Y.H. Therefore it is necessary that the assessors won't be included in the preclinical assessment.

C) Data collection, management and analysis 18. Data collection methods 18.a. Data collection methods: 18.a.i. Baseline data collection: For every patient, medical and dental history will be taken. Examination charts will be filled by M.S.

18.a.ii. Outcome data collection: Modified USPHS criteria for dental restoration will be evaluated by two assessors (M.A & Y.H) at baseline, after 6 ,12 and 18 months, if both assessors differ in score, they will discuss the outcome, if they did not agree, a third assessor (D.M) will resolve the conflict. To achieve inter-examiners reliability, at the beginning of the study, the assessors will perform a profound assessment training program by performing repeated assessments of 36 proximal surface restorations using modified USHPS criteria. The main supervisor (O.S.) will supervise the training program to ensure that the assessors (M.A & Y.H.) will be calibrated before starting their evaluation.

18.b. Patient retention: A record of patient's phone number will be included in every patient's chart. Phone call will be diverted to each patient in order to remind him/her for the time of his/her visit (M.S.). If the patient did not reply for any reason, another visit will be scheduled within a week.

19. Data management: Data entry will be carried out by M.S. and revised by D.M. . All data will be stored on computer and will be encrypted using a password. This will be done to allow accurate data entry through revision and protect data from being incorrectly used. Data will be backed up on another storage device to prevent it from being lost.

20. Statistical methods: Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 25 (SPSS Inc., Chicago, IL).Categorical data will be described as absolute risk for each intervention independently and relative risk when comparing both interventions. Comparisons between categorical variables will be performed using the chi square test. A p-value less than or equal to 0.05 will be considered statistically significant and all tests will be two tailed. Statistical power of the study will be set at 80 % with 95 % confidence level.

D) Data monitoring:

21. Monitoring: The main supervisor (O.S.) will monitor this study. Her role is to monitor any risk of bias could be done from participants, operator or assessors. Also to monitor blinding of the assessors and patient safety, outstanding benefits or harms.

22. Harms: The principle investigator (M.S.) should inform participants about the possible harms (pain, loss of restoration, leakage and fracture of restorations) if present. Participants are allowed to contact the operator at moment through telephone. For assessment radiograph, inspection, percussion and sensitivity tests will be performed. The data will be reported to the co-supervisor (D.M.) and managed through removal of restoration, alleviation of pain and replacement with control restoration.

23. Auditing: In the present trial, auditing will be done by the main supervisors and co-supervisors (O.S. and D.M.) to assure quality of the research methods, restorative technique and interventions.

Section IV:

Ethics and dissemination. 24. Research ethics approval: Application forms for carrying out the clinical trial, checklist and informed consent of Research Ethics Committee (REC) Faculty of Dentistry, Cairo University will be retrieved and filled, then will be delivered for REC committee for approval, this is done to prevent any ethical problems during the study or any harm for any of the participants.

25. Protocol amendments: If a new protocol will be used a protocol amendment will be submitted; containing a new copy of the new protocol and brief explanation about the differences between it and the previous protocols. If there is a change in the existing protocol that affects safety of subjects, investigation scope or scientific quality of the trial, an amendment containing a brief explanation about the change will be submitted. If a new author will be added to accomplish the study, an amendment including the investigator's data and qualifications to conduct the investigation will be submitted to prevent ghost authorship.

26. Consent: Researcher (M.S.) will introduce the trial to patients and provide full explanation of its aim and benefits in plain language. Patients will then be able to have an informed discussion with the researcher. Researcher will obtain written consent from patients willing to participate in the trial. All, consent forms have been translated into Arabic.

27. Confidentiality: Name and personal data of the participants will not appear on the protocol form and will be maintained secured for 10 years after the trial. This is done for protection of participants' privacy and civil rights.

28. Declaration of interests: There is no conflict of interest, no funding or material supplying from any parties.

29. Access to data: Access to final data will be allowed to the operator M.S. and main and co- supervisors (O.S. and D.M.) of the study who are not involved in assessment of the outcome.

30. Ancillary and post-trial care: Patients will be followed up after restoration to ensure oral hygiene measures. When there is any evidence of restoration failure, patients will be treated by immediate restoration removal and control restoration placement.

31. Dissemination policy:

* Full protocol will be published online in Clinicaltrials.gov to avoid repetition, and keep the integrity of the research work.
* Thesis will be discussed and defended in front of a judgment committee.
* The study will be published to report the results of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

-

Patient-related criteria:

* Patients consulting in one of the outpatient clinics listed above.
* Able to tolerate necessary restorative procedures.
* Provide informed consent.
* Accepts the 18 months follow-up period.

Tooth related criteria:

* Teeth with primary proximal carious lesions .
* Teeth are vital according to pulp-sensitivity tests.

Exclusion Criteria:

Patient-related criteria:

* Medically compromised patients, as they will not be able to attend multiple appointments or may require special management.
* Pregnant women; as radiographs cannot be taken for them.
* Allergy to any of the restorative materials, including anesthetics.
* Uncooperative patients, will not abide by the instructions or attend the appointments.

Tooth related criteria:

* Deciduous teeth; as the study is targeting only permanent teeth.
* Teeth with previous restorations, which may add another variable to the study (type of old restorative material, extent of recurrent caries).
* Spontaneous pain or prolonged pain after sensitivity tests (cold and electrical tests), which would indicate irreversible pulpal damage.
* Negative sensitivity tests, periapical radiolucencies and sensitivity to axial or lateral percussion, which would indicate pulp necrosis.
* Teeth presenting external or internal resorption, with adverse pulpal reactions which may affect the outcome of the study.
* Teeth with cervical caries; which can't be evaluated on periapical radiographs.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Fracture | 18 months
  The restoration will be clinically assessed using USPHS criteria. Restorations will be given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.
Marginal adaptation | 18 months
  The restoration will be clinically assessed using USPHS criteria. Restorations will be given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.
Anatomic form | 18 months
  The restoration will be clinically assessed using USPHS criteria. Restorations will be given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.
Surface roughness | 18 months
  The restoration will be clinically assessed using USPHS criteria. Restorations will be given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.
Retention | 18 months
  The restoration will be clinically assessed using USPHS criteria. Restorations will be given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.

SECONDARY OUTCOMES:
Postoperative sensitivity | 18 months
  The restoration will be clinically assessed using USPHS criteria. Restorations will be given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.
secondary caries | 18 months
  The restoration will be clinically assessed using USPHS criteria. Restorations will be given the score Alpha for the ideal clinical situation, Bravo for clinically acceptable and Charlie for clinically unacceptable and in need for replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mohamed sabry Mohamed, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
* Full protocol will be published online in Clinicaltrials.gov to avoid repetition, and keep the integrity of the research work.
  * Thesis will be discussed and defended in front of a judgment committee.
  * The study will be published to report the results of this clinical trial.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 24 months
Access Criteria: open access